CLINICAL TRIAL: NCT03574350
Title: Effect on Early Somatic Growth of a Daily Kinesthetic Stimulation on Preterm Infants Either In Kangaroo Position or in Incubator: A Randomized Control Trial
Brief Title: Effect on Early Somatic Growth of a Daily Kinesthetic Stimulation on Preterm Infants
Acronym: KISONKAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nathalie Charpak (Other)
Collaborators: Laval University (Other); Hospital Universitario San Ignacio (Other)
Responsible Party: Sponsor-Investigator, Nathalie Charpak, Dr Andrea Aldana, Kangaroo Foundation
Organization: Kangaroo Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: KangarooF; xxxxx (Other: Université Laval)
Record Dates: First submitted 2018-06-04; First posted 2018-07-02 (Actual); Last update posted 2018-07-02 (Actual); Status verified 2018-06

CONDITIONS: Preterm Infant; Growth Acceleration; Neurobehavioral Manifestations
Keywords: Kangaroo position; Kinesthetic Stimulation; Kangaroo Mother Care; Bonding
MeSH Terms: conditions — Premature Birth; Neurobehavioral Manifestations | interventions — Incubators

STUDY DESIGN:
Intervention Model Description: Two interventions groups of 33 each, participated in the study. The first group received Kinesthetic Stimulation in Kangaroo Position (KSKP) and the second group received Kinesthetic Stimulation In incubator (KSI ), both of the interventions were delivered by parents during the period of hospitalization and at home when the infant was discharged from Hospital until 40 weeks of gestational age.
Who Masked: Investigator, Outcomes Assessor
Masking Description: The nurses who did anthropometrics measures didn't know the interventions assigned to each participant of the study, because the night shift was in charge of taking the data at 7:00 am in the mornings and the interventions were delivered in the morning shifts from 8:00 am until 5:00 pm. No interventions were delivered in the night.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- KS in Kangaroo Position (KSKP) (Experimental): KS is performed while the infant is in Kangaroo Position using a lycra band to maintain the position.
  Interventions: Behavioral: KS in Kangaroo Position
- KS in incubator (KSI) (Active Comparator): The infant is in the incubator, unclothed with diaper.
  Interventions: Behavioral: KS in incubator

INTERVENTIONS:
Behavioral: KS in Kangaroo Position — KSKP was applied daily at regular interval corresponding to the presence of parents. Our protocol is based on the Tiffany Field's protocol with some adjustments corresponding to the constraints of the hospital : the KS was applied 3 times a day and during 15 consecutive days in the hospital or at home and parents were responsible of delivering the intervention. Sunflower oil was used. During the first 5 days, parents performed KSKP with the support of the psychologist. After day 5, parents were expected to perform KSKP by themselves but could ask for help at any moment while in hospital or in the ambulatory follow-up. The KS always began approximately 60 minutes after the feed.
  Other Names: KSKP
  Arms: KS in Kangaroo Position (KSKP)
Behavioral: KS in incubator — The infant is in the incubator, unclothed with diaper. Parents delivered KSI with the infant in supine position, stroking with the flats of the fingers with moderate pressure. Five 1-minute intervals, consisting of six 10-s periods of stroking, were applied to the following body regions: head, back, both legs and arms. The same process was repeated in prone position. The last part of the intervention was composed of 6 flexions of each extremity.
  Other Names: KSI
  Arms: KS in incubator (KSI)

SUMMARY:
Kangaroo position (KP), the essential component of the Kangaroo Mother Care (KMC) method, has been increasingly implemented, given the benefits of early skin-to-skin contact on the cerebral maturation of preterm infants. In addition it allows for parents to bond with their infants and humanize the care of fragile infants in neonatal units. Evidence on kinesthetic stimulation (KS) is scarce and currently there is no available evidence on KS during the KP. KS is associated with massage in this paper

DETAILED DESCRIPTION:
The objective is to study the impact of standardized KS delivered either in KP (KSKP) or in an incubator (KSI) on the early growth of very preterm infants.

Patients and methods: Sixty six newborns ≤32 weeks of gestational age at birth received KS delivered 3 times/day during KP or in an incubator. They were randomized when the infants were considered eligibleto initiate KMC which was part of the routine care for all newborns in the Neonatal Care Unit (NCU). The primary outcome were the weight gain (g/kg/day) between randomization, 5, and 15 days after the start of the intervention and weight at 40 weeks of gestational age (term). The secondary outcomes were the same measures according to the chronological age (days of life) of the infant at randomization.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infants (GA ≤33 weeks of gestation)
* Deemed clinically stable and eligible for the KMC intervention by the neonatologist were included.

Exclusion Criteria:

* Infants with congenital anomalies
* Unstable during the first 15 days of life

Ages: 30 Weeks to 33 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2013-08-15 (Actual); Primary Completion 2016-08-30 (Actual); Study Completion 2018-02-28 (Actual)

PRIMARY OUTCOMES:
Weight gain after randomization up to 5 days | Between randomization and 5 days post randomization
  weight gain (g/kg/day)
Weight gain after randomization up to 15 days | Between randomization and 15 days post randomization
  weight gain (g/kg/day)
Weight at 40 weeks of gestational age | at 40 weeks of gestational age
  Weight in grames

SECONDARY OUTCOMES:
Weight gain after randomization up to 5 days if randomization was made before 5 days of chronological age | after randomization up to 5 days if randomization was made before 5 days of chronological age
  Weight gain(g/k/d)
Weight gain after randomization up to 15 days if randomization was made before 5 days of chronological age | after randomization up to 15 days of chronological age if randomization was made before 5 days of chronological age
  Weight gain(g/k/d)
Weight at 40 weeks if randomization was made before 5 days of chronological age | at 40 weeks of gestational age if randomization was made before 5 days of chronological age
  Weight in grames
Weight gain after randomization up to 5 days if randomization was made between 6 and 10 days of chronological age | after randomization up to 5 days if randomization was made between 6 and 10 days of chronological age
  Weight gain(g/k/d)
Weight gain after randomization up to 15 days if randomization was made between 6 and 10 days of chronological age | after randomization up to 15 days if randomization was made between 6 and 10 days of chronological age
  Weight gain(g/k/d)
Weight at 40 weeks if randomization was made between 6 and 10 days of chronological age | at 40 weeks of gestational age if randomization was made between 6 and 10 days of chronological age
  Weight in grames
Weight gain after randomization up to 5 days if randomization was made more than 10 days of chronological age | after randomization up to 5 days if randomization was made more than 10 days of chronological age
  Weight gain(g/k/d)
Weight gain after randomization up to 15 days if randomization was made more than 10 days of chronological age | after randomization up to 15 days if randomization was made more than 10 days of chronological age
  Weight gain(g/k/d)
Weight at 40 weeks if randomization was made more than 10 days of chronological age | at 40 weeks of gestational age if randomization was made more than 10 days of chronological age
  Weight in grames

CONTACTS AND LOCATIONS:
Overall Officials: Andrea C Aldana Acosta, PhD, Principal Investigator — Universidad Piloto de Colombia
Locations (1):
- Nathalie Charpak, Bogotá, Cundinamarca, Colombia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Field T, Diego M, Hernandez-Reif M. Potential underlying mechanisms for greater weight gain in massaged preterm infants. Infant Behav Dev. 2011 Jun;34(3):383-9. doi: 10.1016/j.infbeh.2010.12.001. Epub 2011 May 13. PMID 21570125
- [Result] Diego MA, Field T, Hernandez-Reif M. Vagal activity, gastric motility, and weight gain in massaged preterm neonates. J Pediatr. 2005 Jul;147(1):50-5. doi: 10.1016/j.jpeds.2005.02.023. PMID 16027695
- [Result] Guzzetta A, Baldini S, Bancale A, Baroncelli L, Ciucci F, Ghirri P, Putignano E, Sale A, Viegi A, Berardi N, Boldrini A, Cioni G, Maffei L. Massage accelerates brain development and the maturation of visual function. J Neurosci. 2009 May 6;29(18):6042-51. doi: 10.1523/JNEUROSCI.5548-08.2009. PMID 19420271
- See also: Kinesthetic stimulation in Kangaroo Position (KSKP) — https://www.youtube.com/watch?v=WrxDLOBiiZs